CLINICAL TRIAL: NCT00950547
Title: Routinely Use of CardioPAT Cell Saver in Cardiac Surgery: A Prospective Randomized Study Focused on Allogenic Blood Transfusion and Clinical Outcome
Brief Title: ICU Cell Saver to Reduce Blood Transfusions in Cardiac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Saverio Nardella, Cardiochirurgia E.H.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00-02
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Blood Transfusion; Cardiac Surgery
Keywords: Blood Transfusion; Cell Saver; Cardiac Surgery; Evaluate the efficacy of cell salvage CardioPAT routinely used in cardiac surgery in reducing blood transfusions.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Traditional Chest drains
  Interventions: Device: Traditional Chest Drains
- CARDIOPAT (Experimental): CARDIOPAT Cell Saver after Surgery
  Interventions: Device: CARDIOPAT

INTERVENTIONS:
Device: CARDIOPAT — Cell Saver System at bedside for ICU stay
  Arms: CARDIOPAT
Device: Traditional Chest Drains — Chest drains as usual with no possibility to reinfuse lost blood
  Arms: Control

SUMMARY:
PURPOSE: Autotransfusion devices may be employed in cardiac surgery to decrease allogenic blood requirements. Limitations of previous trials include the use of cell saver systems in selected high risk patients only or the lack of blood transfusion-sparing strategies. The aim of this prospective randomized study is to evaluate the efficacy of cell salvage CardioPAT routinely used in cardiac surgery.

METHODS: The investigators will randomize 350 patients in two groups: group 1 receives a CardioPAT cell saver device (175 patients), group 2 doesn't receive any cell saver device. The incidence of allogenic blood transfusion and clinical outcome in both groups are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for cardiac Surgery

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Number of Transfusions per patient | 10 days after surgery

SECONDARY OUTCOMES:
Mortality | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiochirurgia European Hospital, Rome, Italy